CLINICAL TRIAL: NCT02798757
Title: Evaluation of the Tubular Effects of Dapagliflozin Using 1HNMR Spectroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Ass Prof Vasilis Tsimihodimos, Assistant Professor, University of Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10613 - D1690L00044
Record Dates: First submitted 2016-05-30; First posted 2016-06-14 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2017-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapagliflozin (Experimental): All patients will take dapagliflozin, the intervention does not refer to a drug or device but to the specific 1HNMR test spectroscopy
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Urine samples will be collected for 1HNMR spectroscopies

SUMMARY:
This is a phase IV study that will explore the mechanisms of action of a drug (dapagliflozin) that is already commercially available in the country where the study will be conducted (Greece). The drug will be used according to its approved clinical indications (as add-on treatment in patients failed to achieve glycemic targets on metformin monotherapy) and in the approved posology (10 mg/day). Additionally, although there is limited data on the coadministration of dapagliflozin with thiazides, the excellent safety profile of the drug even when it is used in combination with drugs that induce significant volume depletion (such as loop diuretics) suggests that, in properly selected patients, the possibility of important adverse events during the coadministration of dapagliflozin with chlorthalidone is very low. All patients will give written informed consent prior to their enrollment in the study. The study protocol will be approved by the scientific committee of the University Hospital of Ioannina.

DETAILED DESCRIPTION:
Fifty patients with type 2 diabetes on metformin monotherapy with HbA1c > 7% and blood pressure > 140/90 mmHg will be included. All eligible patients will be given dapagliflozin 10 mg qd for 3 months. Routine laboratory parameters that will be measured on each visit include: 1) for serum samples: glucose, urea, creatinine, uric acid, electrolytes (sodium, potassium, chloride, calcium, phosphate and magnesium and 2) for urine samples: glucose, urea, creatinine, uric acid, electrolytes (sodium, potassium, chloride, calcium, phosphate and magnesium) and alpha-1 microglobulin. It is well known that alpha-1 microglobulin is a low-molecular weight protein that is normally filtered by renal glomeruli and reabsorbed by the proximal tubular cells. Increased excretion of alpha1-microglobulin has been proposed as a non-invasive marker for the diagnosis and monitoring of early tubular disorders such as diabetic nephropathy. In addition, the fractional excretion values (FE) of the electrolytes will be calculated using the formula: FEA(%) = (UrineA/SerumA) /(UrineCr/SerumCr) × 100.

The 1HΝMR spectra of urine samples will be recorded on a 500 MHz spectrometer. In the present study, the main low molecular weight (LMW) constituents of urine that will be quantified are 1) metabolites such as glucose, creatinine, creatine, choline, taurine, dimethylamine, betaine, trimethylaminoxide 2) amino acids such as glycine, valine, alanine, leucine, histidine, lysine, threonine and 3) organic acids such as citrate, hippurate, lactate, acetate, succinate, and formate. In addition, 1HNMR methodology allows for the detection of changes in the concentrations of hundreds of metabolites. These substances are normally present in traces, whereas in pathological conditions their concentrations can be found increased.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and/or male aged 18-70 years. Women with childbearing potential can only be included in the study if a serological pregnancy test is negative and a safe contraception method is used throughout the study.
3. Uncontrolled type 2 diabetes mellitus (HbA1c > 7%) on metformin monotherapy (≥ 2000 mg qd or maximum tolerated dose)
4. Stage 1 hypertension (BP 140-159/90-99 mmHg)

Exclusion Criteria:

1. Known primary kidney disease (eGFR < 60 ml/min)
2. History of cardiovascular disease
3. Type 1 diabetes
4. History of heart failure
5. Diseases that shorten the life expectancy (cancers, degenerative neurological disorders etc.)
6. Pregnancy-lactation
7. Patients with eGFR values lower than 45 ml/min (on repeated measurements) during the study period will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Composite outcome measure. % change to the concentrations of specific metabolites. | 6 months
  % change in the concentrations of metabolites such as 1) glucose, creatinine, creatine, choline, taurine, dimethylamine, betaine, trimethylaminoxide 2) amino acids such as glycine, valine, alanine, leucine, histidine, lysine, threonine and 3) organic acids such as citrate, hippurate, lactate, acetate, succinate, and formate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Filippas-Ntekouan S, Dimou A, Dafopoulos P, Kostara C, Bairaktari E, Chasapi S, Spyroulias G, Koufakis T, Koutsovasilis A, Tsimihodimos V. Effect of dapagliflozin on the serum metabolome in patients with type 2 diabetes mellitus. J Diabetes Metab Disord. 2024 Dec 16;24(1):4. doi: 10.1007/s40200-024-01508-1. eCollection 2025 Jun. PMID 39697865
- [Derived] Bletsa E, Filippas-Dekouan S, Kostara C, Dafopoulos P, Dimou A, Pappa E, Chasapi S, Spyroulias G, Koutsovasilis A, Bairaktari E, Ferrannini E, Tsimihodimos V. Effect of Dapagliflozin on Urine Metabolome in Patients with Type 2 Diabetes. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1269-1283. doi: 10.1210/clinem/dgab086. PMID 33592103